CLINICAL TRIAL: NCT03218826
Title: A Phase I Study of AZD8186 in Combination With Docetaxel in Patients With PTEN Mutated or PIK3CB Mutated Advanced Solid Tumors, Potentially Amenable to Docetaxel
Brief Title: PI3Kbeta Inhibitor AZD8186 and Docetaxel in Treating Patients Advanced Solid Tumors With PTEN or PIK3CB Mutations That Are Metastatic or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01232; NCI-2017-01232 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-237; 10131 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10131 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-17 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Prostate Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Castration-Resistant Prostate Carcinoma; Metastatic Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Prostate Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Triple-Negative Breast Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Prostatic Neoplasms; Triple Negative Breast Neoplasms | interventions — Docetaxel; AZD8186

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (docetaxel, PI3Kbeta inhibitor AZD8186) (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 PO BID for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: PI3Kbeta Inhibitor AZD8186

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: PI3Kbeta Inhibitor AZD8186 — Given PO
  Other Names: AZD-8186; AZD8186

SUMMARY:
This phase I trial studies the side effects and best dose of PI3Kbeta inhibitor AZD8186 when given together with docetaxel in treating patients with solid tumors with PTEN or PIK3CB mutations that have spread to other places in the body (metastatic) or cannot be removed by surgery. PI3Kbeta inhibitor AZD8186 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving PI3Kbeta inhibitor AZD8186 and docetaxel may work better in treating patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of PI3Kbeta inhibitor AZD8186 (AZD8186) when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors.

II. To assess the safety and tolerability of AZD8186 when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. Ia. To assess the objective response rate (ORR) of AZD8186 when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors.

Ib. To assess the clinical benefit rate at 24 weeks of AZD8186 when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors.

II. To investigate a drug-drug interaction between docetaxel and AZD8186 and correlate drug exposure with pharmacodynamics response.

EXPLORATORY OBJECTIVES:

I. Examine the pattern of co-mutated genes in PTEN or PIK3CB mutated tumors and their association with treatment response or resistance.

II. Describe possible mechanisms of acquired resistance to PI3Kbeta inhibition. III. Evaluation of protein expression of the PTEN gene and its association with treatment response or resistance.

IV. Examine isoform-specific AKT inhibition and other downstream target modulation from PI3Kbeta inhibition with AZD8186.

OUTLINE: This is a dose-escalation study of PI3Kbeta inhibitor AZD8186.

Patients receive docetaxel intravenously (IV) over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 orally (PO) twice daily (BID) for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must be able to swallow and retain oral medications and be without gastrointestinal illnesses that would preclude absorption of AZD8186
* Unlimited prior therapies allowed
* Docetaxel appropriate

  * Patients who have not received prior docetaxel (or other taxane therapy) in the advanced setting are eligible for all cohorts
  * Patients who have previously received docetaxel (or other taxane therapy) in the advanced setting are eligible for the dose escalation cohort only, if anticipated to have maintained taxane sensitivity and in the opinion of the investigator would still benefit from further docetaxel therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 8 g/L
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* PTEN or PIK3CB mutated advanced solid tumor

  * PTEN loss of function mutation or PIK3CB gain of function mutation identified by local Clinical Laboratory Improvement Act (CLIA) certified next generation sequencing (NGS)
  * Breast cancers patients enrolled on this study must have either:

    * Estrogen receptor positive and HER2 negative breast cancer
    * Triple negative breast cancer
* Adequate archival tissue (metastatic tissue sample is preferable but primary tumor tissue will be acceptable) or willing to undergo pre-treatment biopsy (for central confirmation of molecular alteration and PTEN immunohistochemical assessment) if adequate archival tissue is unavailable
* The effects of AZD8186 on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of AZD8186 administration
* Ability to understand and the willingness to sign a written informed consent document
* DOSE ESCALATION COHORT: Prior receipt of docetaxel is permitted
* DOSE ESCALATION COHORT: Measurable disease is not required for enrollment
* PHARMACODYNAMIC EXPANSION COHORT: Prior receipt of docetaxel is not permitted
* PHARMACODYNAMIC EXPANSION COHORT: Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* PHARMACODYNAMIC EXPANSION COHORT: Consent to allow mandatory paired (pre- and on- treatment) fresh tissue biopsies if deemed safe to do so for quantitation of Akt pathway signaling proteins
* DISEASE SPECIFIC EXPANSION COHORTS: Prior receipt of docetaxel is not permitted
* DISEASE SPECIFIC EXPANSION COHORTS: Patients (excepting the prostate cancer patients) must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* DISEASE SPECIFIC EXPANSION COHORTS: Breast cancers patients enrolled on this study must have:

  * Metastatic or advanced (incurable and unresectable) HER2 negative breast cancer regardless of estrogen receptor status (both hormone receptor positive and triple negative patients are eligible)
  * Received hormonal therapy, as appropriate based on their hormone receptor status; hormone receptor positive patients who have not received endocrine therapy for recurrent/metastatic disease are eligible, permitted their physician feels they are not appropriate for first line endocrine therapy, for example for high risk visceral metastatic disease
* DISEASE SPECIFIC EXPANSION COHORTS: Prostate cancers patients enrolled on this study (applies to all prostate cancer patients treated on parts 1, 2, and 3) must have:

  * Metastatic or advanced (incurable and unresectable) castration resistant metastatic cancer
  * Received at least one additional line of anti-androgen therapy with abiraterone or enzalutamide
  * Measurable disease is not required for enrollment

Exclusion Criteria:

* HER2 positive breast cancer
* Prior treatment with PI3K/AKT inhibitors
* Any known concurrent RAF or PIK3CA mutation
* Patients who have had chemotherapy, radiotherapy, immunotherapy or anticancer agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of the first dose of study treatment, except hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with prostate cancer and breast cancer, which are permitted
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* Patients with known, untreated or unstable brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients with treated brain metastases are eligible if the metastases have been radiographically and clinically stable for at least one month; if on steroids for this indication, the patient must be on a stable dose for at least one month
* History of clinically significant allergic reactions attributed to compounds of similar chemical or biologic composition to AZD8186 or docetaxel or to docetaxel itself
* Patients receiving any medications or substances that are strong inhibitors and/or strong or moderate inducers of CYP3A4 are ineligible; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Existing bleeding or condition associated with increased risk of bleeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD8186 is a PI3K inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD8186, breastfeeding should be discontinued if the mother is treated with AZD8186; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART) that does not include strong inhibitors and strong or moderate inducers of CYP3A4
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2026-10-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Schram, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (8):
- United States (8):
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Schram AM, Takebe N, Chen A, Zhou Q, Iasonos A, Silber J, Reynolds M, Hussain S, Gavriliuc M, Smyth LM, Garrison D, Dumbrava EE. A phase I study of AZD8186 in combination with docetaxel in patients with PTEN-mutated or PIK3CB-mutated advanced solid tumors. ESMO Open. 2025 Sep;10(9):105569. doi: 10.1016/j.esmoop.2025.105569. Epub 2025 Sep 11. PMID 40939237
- [Derived] Schrottmaier WC, Kral-Pointner JB, Salzmann M, Mussbacher M, Schmuckenschlager A, Pirabe A, Brunnthaler L, Kuttke M, Maier B, Heber S, Datler H, Ekici Y, Niederreiter B, Heber U, Blomgren B, Gorki AD, Soderberg-Naucler C, Payrastre B, Gratacap MP, Knapp S, Schabbauer G, Assinger A. Platelet p110beta mediates platelet-leukocyte interaction and curtails bacterial dissemination in pneumococcal pneumonia. Cell Rep. 2022 Nov 8;41(6):111614. doi: 10.1016/j.celrep.2022.111614. PMID 36351402

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1; Dose Level 1 With Growth Factors: Patients receive docetaxel 75 mg/m^2 IV over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 60 mg PO BID for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.
- Dose Level -1: Patients receive docetaxel 75 mg/m^2 IV over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 30 mg PO BID for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.
- Dose Level -1B: Patients receive docetaxel 60 mg/m^2 IV over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 60 mg PO BID for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.
- Dose Level 2: Patients receive docetaxel 75 mg/m^2 IV over 1 hour on day 1 and PI3Kbeta inhibitor AZD8186 120 mg PO BID for 5 days each week. Cycles repeat every 21 days until April 30, 2022 in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Started | 6 | 1 | 5 | 4 | 7
Completed | 5 | 1 | 3 | 3 | 6
Not Completed | 1 | 0 | 2 | 1 | 1
Not completed — Non-compliance with protocol | 1 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2 | Total
Number analyzed (Participants) | 6 | 1 | 5 | 4 | 7 | 23
Age, Continuous [Median (Full Range); unit: years] | 50 [40 to 74] | 56 [56 to 56] | 55 [38 to 76] | 56 [49 to 63] | 61 [36 to 80] | 56 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 4 | 3 | 16
  Male | 2 | 0 | 1 | 0 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 1 | 4 | 4 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 5 | 1 | 5 | 3 | 7 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 5 | 4 | 7 | 23
Height [Median (Full Range); unit: centimeter (cm)] | 168.5 [156.5 to 176] | 183 [183 to 183] | 170 [150 to 177] | 160.5 [155 to 165.1] | 170 [159 to 189] | 168 [150 to 189]
Weight [Median (Full Range); unit: kilogram (kg)] | 79.5 [62.6 to 94] | 100 [100 to 100] | 58.6 [54.7 to 79.5] | 68 [44.4 to 115.2] | 77.9 [61.5 to 111.3] | 76.2 [44.4 to 115.2]
Body Surface Area [Median (Full Range); unit: meters squared (m^2)] | 1.86 [1.75 to 2.07] | 2.22 [2.22 to 2.22] | 1.68 [1.51 to 1.95] | 1.73 [1.38 to 2.19] | 1.94 [1.69 to 2.42] | 1.90 [1.38 to 2.42]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: The number of DLTs at each dose level will determine the MTD or RP2D of PI3Kbeta inhibitor AZD8186 when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors.
Time Frame: At Day 22
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 6
Participants
  Experienced Dose Limiting Toxicity | 2 | 0 | 0 | 0 | 0
  Did not experience Dose Limiting Toxicity | 3 | 1 | 3 | 3 | 6

2. Primary Outcome: Number of Participants With Adverse Events (AEs) Grades 3-5
Description: Patient safety and tolerability will be described according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version for routine toxicity reporting and CTCAE, version 5 for serious adverse events only.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 6
Participants
  Experienced AEs grades 3-5 | 4 | 1 | 3 | 1 | 4
  Not Experienced AEs grades 3-5 | 1 | 0 | 0 | 2 | 2

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR. For participants with prostate cancer who do not have sites of disease on imaging, objective response is the reduction of prostate specific antigen (PSA) level of 50% or more.
Time Frame: At 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 6
Participants
  Objective response | 0 | 0 | 1 | 0 | 0
  No objective response | 5 | 0 | 2 | 2 | 5
  Not assessed | 0 | 1 | 0 | 1 | 1

4. Secondary Outcome: Clinical Benefit Rate (CBR) Defined as Complete Response (CR), Partial Response (PR), or Stable Disease
Description: Will be assessed by modified Response Evaluation Criteria in Solid Tumors version 1.1. Will assess the CBR of PI3Kbeta inhibitor AZD8186 when administered in combination with docetaxel in patients with PTEN or PIK3CB mutated advanced solid tumors. A 90% confidence interval on CBR will be calculated assuming binomial proportions.
Time Frame: At 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 6
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 1 | 0 | 0
  Stable Disease (SD) | 1 | 0 | 0 | 0 | 1
  Progressive Disease (PD) | 4 | 0 | 2 | 2 | 4
  Not assessed | 0 | 1 | 0 | 1 | 1

5. Secondary Outcome: Maximum Blood Concentrations of Docetaxel When Also Taking AZD8186
Description: Will investigate the concentration of docetaxel in the blood when participants also take the PI3Kbeta inhibitor AZD8186. Blood is drawn after docetaxel infusion and before the participant takes AZD8186, after the participant takes AZD8186, and again 6 hours after taking AZD8186. Blood concentrations of docetaxel are measured at each collection time. The change in concentrations at the different dose levels may suggest whether AZD8186 impacts how much docetaxel is still in the blood over time.
Time Frame: Up to 6 hours after initial treatment
Population: Test not collected for pts on dose level -1.
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
Number analyzed (Participants) | 3 | 0 | 1 | 3 | 6
ng/ml
  Pre-Treatment | 3083.3 (1933.8) |  | 2060.0 (0) | 3280.0 (585.1) | 3450.0 (1735.9)
  After Treatment: number analyzed (Participants) | 3 | 0 | 1 | 1 | 6
  After Treatment | 6981.7 (4457.9) |  | 3615.0 (0) | 4728.6 (0) | 6493.9 (3437.8)
  6 Hours after Treatment: number analyzed (Participants) | 3 | 0 | 1 | 1 | 6
  6 Hours after Treatment | 6213.8 (3991.4) |  | 3056.1 (0) | 4411.6 (0) | 7008.0 (3877.0)

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -1B | Dose Level 1 With Growth Factors | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 4/6 | 1/1 | 3/5 | 2/4 | 2/7
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/1 | 4/5 | 1/4 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1 | 5/5 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level -1 (N=1) | Dose Level -1B (N=5) | Dose Level 1 With Growth Factors (N=4) | Dose Level 2 (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 2 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level -1 (N=1) | Dose Level -1B (N=5) | Dose Level 1 With Growth Factors (N=4) | Dose Level 2 (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1
Alkaline phosphatase increased (Investigations) | 3 | 0 | 2 | 2 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 3
ALT level increased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 2 | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Eye twitching (Eye disorders) | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 1 | 2 | 3
Fever (General disorders) | 0 | 0 | 1 | 0 | 1
Finger Cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 2
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 3 | 1 | 3
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nail Lifting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 4
Neutrophil count decreased (Investigations) | 2 | 0 | 3 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Prolapsed Bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Root canal procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Thrush (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Toe nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tooth pain / Swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1 | 1 | 0
White blood cell decreased (Investigations) | 2 | 1 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03218826/Prot_SAP_000.pdf